CLINICAL TRIAL: NCT04319887
Title: A Prospective, Multicenter, Single-arm Study Examining ECAP-controlled, Closed-loop Stimulation With the Evoke Spinal Cord Stimulator (SCS) System to Treat Patients With Chronic Pain of the Trunk and/or Limbs
Brief Title: ECAP-controlled, Closed-loop Stimulation to Treat Chronic Trunk and/or Limb Pain (ECAP)
Acronym: ECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-PCL-006732
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain; Back Pain; Pain
Keywords: Chronic Pain; Back Pain; Leg Pain; Pain; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; SCS; Closed Loop
MeSH Terms: conditions — Chronic Pain; Back Pain; Pain; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ECAP-controlled, closed-loop SCS (Experimental): Spinal cord stimulation that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude
  Interventions: Device: Evoke Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Evoke Spinal Cord Stimulation (SCS) System — A spinal cord stimulation system that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude

SUMMARY:
The purpose of this study is to evaluate neurophysiological measures and clinical outcomes of the Evoke System to treat trunk and/or limb pain in a real-world population.

ELIGIBILITY:
Inclusion Criteria:

* Subject has chronic intractable pain of the trunk and/or limbs.
* Subject is willing and capable of giving informed consent and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

* Subject is unable to operate the system.
* Subject is an unsuitable surgical candidate.
* Subject has a condition currently requiring or likely to require the use of diathermy.
* Subject has another implantable stimulator such as demand type pacemakers or cardioverter defibrillator.
* Subject is <18 years old.
* Subject is pregnant or nursing.
* Subject is allergic, or has shown hypersensitivity, to any materials of the neurostimulation system which come in contact with the body.
* Subject is being treated with electroconvulsive therapy (ECT) or transcranial magnetic stimulation (rTMS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - Pacific Research Institute, Santa Rosa, California
  - The Orthopaedic Institute, PA, Gainesville, Florida
  - Alliance Spine and Pain Centers, Atlanta, Georgia
  - Southern Pain and Spine, Fayetteville, Georgia
  - Axis Spine Center, Hayden Lake, Idaho
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Ochsner Clinic, New Orleans, Louisiana
  - Interventional Spine and Pain Physicians, Maple Grove, Minnesota
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Albany Medical College, Albany, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Spinal Diagnostics, PC, Tualatin, Oregon
  - Delaware Valley Pain & Spine Institute, Feasterville-Trevose, Pennsylvania
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - Sprintz Center for Pain PLLC, Shenandoah, Texas
  - Precision Spine Care, Tyler, Texas
  - St. Francis Hospital, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pope JE, Antony A, Petersen EA, Rosen SM, Sayed D, Hunter CW, Goree JH, Vu CM, Bhandal HS, Shumsky PM, Bromberg TA, Smith GL, Lam CM, Kalia H, Lee JM, Khurram A, Gould I, Karantonis DM, Deer TR. Identifying SCS Trial Responders Immediately After Postoperative Programming with ECAP Dose-Controlled Closed-Loop Therapy. Pain Ther. 2024 Oct;13(5):1173-1185. doi: 10.1007/s40122-024-00631-4. Epub 2024 Jul 9. PMID 38977651

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single-arm study. Subjects undergo a trial with the device, at which point they are enrolled, prior to receiving a permanent implant. Results are for implanted subjects.
Period: Overall Study
Arm/Group | ECAP-controlled, Closed-loop SCS
Started | 231
Completed | 208
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | ECAP-controlled, Closed-loop SCS
Number analyzed (Participants) | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 218
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 217
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 231

OUTCOME MEASURES:

1. Primary Outcome: Evoked Compound Action Potentials (ECAPs) as Measured by the Evoke SCS System
Description: Dose ratio is determined by the estimated current (mA) at the median ECAP level divided by the current (mA) at the ECAP threshold. The dose ratio allows for both the individualization of a patient's neural dose and comparison across patients, using their ECAP threshold and unique dose response. This metric normalizes for distance between the electrode and the spinal cord and the distances between the stimulation and recording electrodes. The dose ratio reflects the amount of dorsal column activation elicited by stimulation with respect to threshold levels. For example, if the dose is at ECAP threshold, this value will be 1. If the dose is 30% higher than ECAP threshold, this value will be 1.3.
Time Frame: 12-months post-implant
Population: patients who completed the 12-month follow-up visit
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | ECAP-controlled, Closed-loop SCS
Number analyzed (Participants) | 208
ratio | 1.3 [1.1 to 1.5]
Statistical Analysis 1: Comparison: ECAP-controlled, Closed-loop SCS; Test type: Other; statistical analysis section may be deleted

2. Other Pre Specified Outcome: Change in Pain
Description: Visual Analogue Scale (VAS) to rate pain intensity
Time Frame: end of trial period; 1-, 3-, 6-, 12-, 18-, and 24-months post-implant
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in PROMIS-29
Description: 29-item profile instrument that assesses 8 universal domains (not disease-specific): Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity.
Time Frame: end of trial period; 1-, 3-, 6-, 12-, 18-, and 24-months post-implant
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in PROMIS-10 Global
Description: 10-item instrument that assesses Physical Health and Mental Health
Time Frame: end of trial period; 1-, 3-, 6-, 12-, 18-, and 24-months post-implant
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Profile of Mood States (POMS 2-A Short)
Description: 35-item instrument that assesses mood states overall (Total Mood Disturbance) and six mood clusters: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. A scale score is also calculated for Friendliness.
Time Frame: end of trial period; 1-, 3-, 6-, 12-, 18-, and 24-months post-implant
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Rate of Patient Global Impression of Change (PGIC)
Description: Single item measure of global improvement with treatment
Time Frame: end of trial period; 1-, 3-, 6-, 12-, 18-, and 24-months post-implant
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Rate of Patient Satisfaction With Therapy
Description: Single item measure of satisfaction with treatment
Time Frame: end of trial period; 1-, 3-, 6-, 12-, 18-, and 24-months post-implant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE data were collected from consent through study completion/exit, an average of 1 year.
Description: SAE criteria:
  * Led to death,
  * Led to serious deterioration in the health of the subject, and that either resulted in:
    1. a life-threatening illness or injury, or
    2. a permanent impairment of a body structure or a body function, or
    3. prolonged hospitalization, or
    4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
  * Led to fetal distress, fetal death, or congenital anomaly or birth defect.
Arm/Group | ECAP-controlled, Closed-loop SCS
All-Cause Mortality (participants affected / at risk) | 3/300
Serious Adverse Events (participants affected / at risk) | 38/300
Other Adverse Events (participants affected / at risk) | 59/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECAP-controlled, Closed-loop SCS (N=300)
Fall or Trip or Slip or Twist (Injury, poisoning and procedural complications) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3)
Cholelithiasis or Gallstones (Hepatobiliary disorders) | 2 (2)
Dural Puncture or Tear (Nervous system disorders) | 2 (2)
Nerve Root or Spinal Cord Injury (Nervous system disorders) | 2 (2)
Overdose (Psychiatric disorders) | 2 (2)
Septicemia (Infections and infestations) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Activities of Daily Living (ADL) Injury (Injury, poisoning and procedural complications) | 1 (1)
Allergic Reaction - Medications or Dressings (Immune system disorders) | 1 (1)
Arrhythmia and Irregularities (Cardiac disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Autoimmune, non-specific (Immune system disorders) | 1 (1)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain Hemorrhage (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Coronary Artery or Heart Disease (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Disorientation (Nervous system disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Hematoma (Immune system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inflammation (Endocrine disorders) | 1 (1)
Kidney Problems - Other (Renal and urinary disorders) | 1 (1)
MRSA (Infections and infestations) | 1 (1)
Myocardial Infarct or Heart Attack (Cardiac disorders) | 1 (1)
Non-specific Infection (Immune system disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper Respiratory Symptoms or Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound Dehiscence (Immune system disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECAP-controlled, Closed-loop SCS (N=300)
Fall or Trip or Slip or Twist (Injury, poisoning and procedural complications) | 37 (42)
Upper Respiratory Symptoms or Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Activities of Daily Living (ADL) Injury (Injury, poisoning and procedural complications) | 16 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish their site's results if:

* Multi-center results are published, unless authorized by Sponsor. If multi-center results are not submitted within 12 months of clinical trial conclusion, PI may publish their results; AND
* Provide Sponsor 60 days to review. If Sponsor response not received within 60 days, PI may publish. If Sponsor determines the proposed publication contains confidential or patentable information, Sponsor may delay publication for up to 90 days from discovery.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT04319887/Prot_SAP_001.pdf